CLINICAL TRIAL: NCT04945668
Title: Combined Ultrasound and Fluoroscopy-guided Technique for Treatment of Hip Pain. A Pilot Study for a Suggested Approach for Anterior Hip Denervation
Brief Title: Combined Ultrasound and Fluoroscopy-guided Technique for Anterior Hip Denervation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MFM-IRB, R.21.05.1337
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pericapsular nerve group block (Other): combined ultrasound and fluoroscopy-guided technique for pericapsular nerve group block
  Interventions: Procedure: Modified technique for pericapsular nerve group block

INTERVENTIONS:
Procedure: Modified technique for pericapsular nerve group block — with the patient in the supine position, ultrasound probe in a transverse plane over the anterior inferior iliac spine (AIIS) and then aligned with the pubic ramus. In this view, the ilio pubic eminence (IPE), the iliopsoas muscle and tendon will be observed. A spinal needle will be inserted from lateral to medial in an in-plane approach to place the tip between the psoas tendon and the pubic ramus. Fluoroscopic image will be taken to confirm the needle tip position in the target site. Following negative aspiration, 15 ml dye will be injected in 5-mL increments while observing for adequate spread using fluoroscopy followed by 15ml local anesthetic

SUMMARY:
Hip fracture is a challenging geriatric problem for health care professionals, especially in patients with multiple comorbidities. In patients with inoperable hip fractures secondary to severe comorbid conditions, the pain can lead to significant challenges in nursing care.

A recent anatomical study confirmed the innervation of the anterior hip by these 3 main nerves but also found that the AON and FN play a greater role in the anterior hip innervation than previously reported.

DETAILED DESCRIPTION:
The aim of this study is to help to target a suggested optimum landmark and determine the volume of injectate that can cover the distribution of the anterior articular branches supplying the hip joint.

The anterior hip capsule is innervated by the ON, accessory obturator nerve (AON), and FN as reported by previous anatomic studies. The anterior capsule is the most richly innervated section of the joint.

Ultrasound-guided technique for blockade of these articular branches to the hip, the PENG (Pericapsular Nerve Group) block reported significantly reduced pain scores compared with baseline.

With the current understanding of the complex innervations of the hip joint, it is difficult to provide complete effective radiofrequency ablation to the articular branches supplying the hip joint. Chemical hip denervation using ultrasound was reported by previous case reports or series without mentioning a well-defined target point or an optimum injectate volume.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II, and III.
* Patients scheduled for elective or emergent hip fractures.

Exclusion Criteria:

* Patient refusal.
* Neuromuscular diseases (as myopathies, myasthenia gravies…)
* Hematological diseases, bleeding, or coagulation abnormality.
* Psychiatric diseases.
* Local skin infection and sepsis at the site of the block.
* Known intolerance to the study drugs.
* Body Mass Index > 40 Kg/m2.
* Multiple trauma patients.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The success rate to target a suggested optimal landmark | just after skin puncture
  Is defined as the percentage of success to reach the target point for injection with needle punctures to up to 4 skin punctures.

SECONDARY OUTCOMES:
Success rate of first skin puncture | just after skin puncture
  Is defined as the number of getting the target point from the first skin puncture
The number of skin punctures: | just after skin puncture for the block
  Is defined as the total number of skin punctures for either getting the target point or not.
the total number of needle passes required for obtaining the target landmark | just after skin puncture
  Is defined as the total number of forward advancements of the spinal needle i.e. withdrawal and redirection without exiting the skin (sum of passes of all punctures).
The optimum volume of the injectate | 30 minutes before surgery.
  Is defined as the optimum volume of the injectate to cover the target innervation area.
Pain measurement at rest | Prior to performing of nerve block, 15, 30 minutes after block performance
  10-cm visual analog scale (VAS) for pain, where 0 is equal to no pain and 10 indicates the worst possible pain.
Pain measurement on movement (attempted hip flexion to 15 degrees): | Prior to performing of nerve block, 15, 30 minutes after block performance
  10-cm visual analog scale (VAS) for pain, where 0 is equal to no pain and 10 indicates the worst possible pain,
Incidence of block failed block | 30 minutes after Local Anesthetic injection
  Is defined as less than 50% pain relief of pain i.e. (less than 50% of VAS score is reduced after the block
Time for first analgesic request | Within 24 hours after surgery
  the time passed from LA injection to the patient need of first analgesia
Patient satisfaction score | Within 24 hours after the nerve block
  From zero=Poor, 1=fair, 2=good, 3=very good to 5=excellent
Complications: | Within 24 hours after the nerve block
  presence or absence of unintentional vascular puncture, hematoma formation, parasthesia

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Y Makharita, M.D., Study Chair — Professor of Anesthesia and Surgical Intensive Care; Shimaa Shalaby, M.Sec., Principal Investigator — Assistant lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after completing the study and being accepted for publication.
Access Criteria: The data will be accessible to the investigators and PRS administrators with hiding the identifiers for the patients